CLINICAL TRIAL: NCT01748669
Title: Effectiveness of Garlic Oil in the Treatment of Arsenical Palmer Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Prof. Mir Misbahuddin, Prof. and Chairman, Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU-005-CT
Record Dates: First submitted 2012-12-11; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Arsenic Poisoning
Keywords: Arsenic; Arsenicosis; Garlic oil; Keratosis
MeSH Terms: conditions — Keratosis | interventions — allyl sulfide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients of palmer arsenical keratosis (Experimental): One soft capsule of garlic oil (10 mg) daily for 12 weeks
  Interventions: Dietary Supplement: Garlic oil
- Arsenic exposed controls (Active Comparator): One soft capsule of garlic oil (10 mg) daily for 12 weeks
  Interventions: Dietary Supplement: Garlic oil
- Heathy volunteers (Active Comparator): One soft capsule of garlic oil (10 mg) daily for 12 weeks
  Interventions: Dietary Supplement: Garlic oil

INTERVENTIONS:
Dietary Supplement: Garlic oil — Oral administration

SUMMARY:
Twenty patients of mild to moderate degree of arsenical palmer keratosis will be treated with garlic oil capsule orally for 12 weeks to examine its effectiveness in reducing body arsenic load and clinical symptoms. Similar treatment with similar number of arsenic exposed controls and healthy volunteers will be included for comparison.

DETAILED DESCRIPTION:
Thousands of Bangladeshi are suffering from arsenic-induced keratosis affecting palms and soles. Palmer keratosis, particularly in young female, affects the socioeconomic condition. Till today there is no effective treatment.

Twenty patients of mild to moderate degree of arsenical palmer keratosis will be treated with garlic oil in soft capsule (10 mg/day) orally for 12 weeks. Similar treatment will be given to 20 arsenic exposed controls and 20 healthy volunteers for comparison. The aim of this study is to examine the effectiveness of oral administration of garlic oil to reduce body arsenic load and clinical symptoms of arsenical palmer keratosis.

ELIGIBILITY:
Inclusion Criteria (Patients):

* history of taking arsenic contaminated water (>50 ppb) for more than 6 months
* patients having mild to moderate arsenical keratosis present on palm of the hand
* patients those voluntarily agree to participate

Inclusion Criteria (Arsenic exposed controls):

* family member of the patient
* drinking arsenic contaminated water from the same source as patient
* those voluntarily agree to participate
* no sign/symptom of palmer keratosis

Inclusion Criteria (Healthy volunteers):

* drinking arsenic safe water (<50 ppb)
* those voluntarily agree to participate

Exclusion Criteria:

* pregnancy
* lactating mother
* patient receiving treatment of arsenicosis
* any other chronic disease like tuberculosis, diabetes mellitus, bronchial asthma

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in the clinical symptom of keratosis in palm | 0 week (baseline) to 12 weeks (end)

SECONDARY OUTCOMES:
Change in biochemical parameters (blood sugar, cholesterol and transaminase) after treatment | 0 week (baseline), 12 weeks (end)
Adverse effects following treament | 0 week (baseline), 12 weeks (end)
Change in the amount of arsenic in nail | 0 week (baseline), 20 weeks (end)

CONTACTS AND LOCATIONS:
Overall Officials: Mir Misbahuddin, MBBS, PhD, Principal Investigator — Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh.
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh